CLINICAL TRIAL: NCT07190300
Title: TulmiSTAR-02: A Two-part Phase I Dose Escalation Study of Tulmimetostat (DZR123) in Combination With Darolutamide or Abiraterone Followed by Open-label, Randomized, Phase II Dose Expansion Study to Assess the Safety and Efficacy of Tulmimetostat in Combination With Darolutamide Versus Darolutamide Alone in Patients With Metastatic Hormone-sensitive Prostate Cancer
Brief Title: TulmiSTAR-02: A Phase I/II Open-label Study of Tulmimetostat in Combination With Darolutamide vs. Darolutamide, and Tulmimetostat With Abiraterone in Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Acronym: TulmiSTAR-02
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDZR123C12101; 2025-521873-15-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC); Enhancer of Zeste Homolog 2 (EZH2); Androgen Receptor (AR); Androgen Receptor Pathway Inhibitors (ARPIs); Prostate-Specific Antigen (PSA); Biochemical Response Rate (BCR); TulmiSTAR-02
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — darolutamide; abiraterone

STUDY DESIGN:
Intervention Model Description: Phase I (Part 1 and Part 2) = Open-label Phase II = Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I: Group A (part 1) (Experimental): Tulmimetostat oral (PO) once a day (QD) escalating doses + Darolutamide 600 mg twice a day (BID)
  Interventions: Drug: Tulmimetostat; Drug: Darolutamide
- Phase I: Group B (part 2) (Experimental): Tulmimetostat PO QD escalating doses + Abiraterone 1000 mg PO QD
  Interventions: Drug: Tulmimetostat; Drug: Abiraterone
- Phase II: Arm 1 (Experimental): Tulmimetostat dose 1 PO + Darolutamide 600 mg PO BID
  Interventions: Drug: Tulmimetostat; Drug: Darolutamide
- Phase II: Arm 2 (Experimental): Tulmimetostat dose 2 PO + Darolutamide 600 mg PO BID
  Interventions: Drug: Tulmimetostat; Drug: Darolutamide
- Phase II: Arm 3 (Active Comparator): Darolutamide 600 mg PO BID
  Interventions: Drug: Darolutamide

INTERVENTIONS:
Drug: Tulmimetostat — Doses of tulmimetostat beyond DL1 once a day (QD) will be opened depending on outcome of Dose Escalation Meetings (DEM(s))
  Other Names: DZR123
  Arms: Phase I: Group A (part 1); Phase I: Group B (part 2); Phase II: Arm 1; Phase II: Arm 2
Drug: Darolutamide — 600 mg is administered orally BID
  Arms: Phase I: Group A (part 1); Phase II: Arm 1; Phase II: Arm 2; Phase II: Arm 3
Drug: Abiraterone — abiraterone 1000 mg is administered orally QD
  Arms: Phase I: Group B (part 2)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and efficacy of the two different treatment combinations of tulmimetostat in participants with de novo or recurrent Metastatic Hormone-Sensitive Prostate Cancer (mHSPC).

DETAILED DESCRIPTION:
The study consists of two phases:

1. The Phase I part includes two groups: Part 1 will assess the combination of tulmimetostat with darolutamide (Group A), and Part 2 will assess tulmimetostat with abiraterone (Group B). The primary objective of Phase I is to determine the Recommended Dose Escalations (RDEs) for each combination, with enrollment using a staggered approach between the groups. Participants in both Group A and Group B will continue androgen deprivation therapy (ADT) to maintain castrate testosterone levels (< 50 ng/dL or < 1.7 nmol/L), with the ADT modality determined by the investigator based on local guidelines. In Group B, abiraterone will be co-administered with an oral corticosteroid (prednisone or prednisolone) as per local prescribing information.
2. The Phase II part is a randomized, open-label, multicenter dose-expansion study designed to further evaluate the recommended dose(s) of tulmimetostat in combination with darolutamide and provide proof-of-concept for its efficacy and safety. Participants in Phase II will be randomized to receive either tulmimetostat plus darolutamide or darolutamide alone. Eligible participants include those with de novo or recurrent mHSPC who have not previously received prior radioligand therapy but may have prior exposure to taxane-based chemotherapy and/or androgen receptor pathway inhibitors (ARPI, excluding darolutamide). This study aims to explore tulmimetostat-based combinations as potential therapeutic options for men with mHSPC.

The study for each participant consists of a screening period, a study treatment period followed by a post treatment long-term follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult men ≥ 18 years old with de novo or recurrent mHSPC (without neuroendocrine or small cell features). The tumor lesion(s) may be located in the bone, soft tissue/visceral region, or both.
* Participants must have castrate levels of testosterone, i.e., ≤ 50 ng/dL (≤ 1.7 nM).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Adequate bone marrow and organ function
* Prior ADT: Participants must have started ADT at least 1 month but no more than 24 months before study entry and be willing to continue ADT during treatment
* Prior taxane use for mHSPC:

  ~ Phase I and II: Participants may have received, but not progressed on, one prior taxane-based therapy. Phase II: Limited to 25% participants with prior taxane use.
* Prior ARPI (abiraterone, enzalutamide, darolutamide, or apalutamide) is allowed in both Phase I and Phase II:

  1. Prior ARPI use in biochemical recurrence (BCR) or curative treatment is allowed for any duration, provided therapy was discontinued and participant had no evidence of conventional imaging positive metastatic disease at that time
  2. Prior ARPI use in mHSPC

     * Phase I: Allowed for any duration.
     * Phase II: Allowed prior exposure to ARPI is ≤6 months. Participants with ongoing use of darolutamide are not eligible.

     Note: Participants are required to stop their prior ARPI after providing their consent to join this study. Participants with ongoing ARPI are eligible for a switch from their ongoing ARPI therapy if they have not progressed to CRPC disease, and meet any of the criteria, indicative of suboptimal biochemical response, or intolerability, as assessed by the Investigator.
* Other permitted prior local therapy for mHSPC:

  * Phase I and II: Prior prostate-directed radiation or surgical intervention. Radiation must be completed before study entry; surgery at least 2 weeks prior.

Key Exclusion Criteria:

* Participants with evidence of mCRPC or biochemical recurrence / PSA only disease or asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy and with normal PSA for ≥ 1 year prior to the start of study treatment.
* Participants with PSA levels of ≤ 0.2 ng/mL at the start of study treatment.
* Participants with CNS metastases are excluded unless:

  * they have received prior therapy (e.g. surgery, radiotherapy, gamma knife), are neurologically stable and asymptomatic
  * they are not receiving corticosteroid for the purpose of maintaining neurologic integrity and have baseline and subsequent radiological imaging of the brain.
  * Participants with epidural disease, canal disease, or prior spinal cord involvement are excluded unless these areas have been treated, are stable, and the participant is not neurologically impaired.
* Concurrent use of first-generation anti-androgens (like bicalutamide). Prior use of a first-generation anti-androgen drug in the context of ADT initiation with a GNRH analog is allowed, provided it was administered for ≤14 days and the last dose was administered ≥7 days from the study entry.
* Systemic ketoconazole is used as antineoplastic treatment for prostate cancer.
* Previous exposure to radioligand therapy.
* Treatment with any investigational agent within 28 days (or 5 half-lives, whichever is longer) prior to study entry.
* Previous treatment with any Polycomb Repressive Complex 2 (PRC2) inhibitor, including but not limited to Enhancer of Zeste Homolog 2 (EZH2) inhibitors, EZH2/1 inhibitors, or embryonic ectoderm development (EED) inhibitors.
* Herbal products that may decrease PSA levels within 4 weeks prior to the start of study drug treatment and while on study
* Participants taking prohibited medication(s) (e.g., strong CYP3A4 inducers or strong or moderate CYP3A4 inhibitors that cannot be stopped within 7 days or 5 half-lives (whichever is longer) prior to study treatment and for the duration of the study treatment or prohibited herbal product(s) that cannot be stopped 7 days prior to study treatment.

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2032-06-04 (Estimated); Study Completion 2032-06-04 (Estimated)

PRIMARY OUTCOMES:
Phase I (Group A and Group B): Dose-limiting toxicities (DLTs) | Up to 28 days
  A dose-limiting toxicity is defined as an adverse event or abnormal laboratory value, not clearly due to underlying disease or extraneous causes, that occurs within the first 28 days of treatment with tulmimetostat and meets any of the criteria specified in the protocol. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for all grading. For the purpose of dose-escalation decisions, DLTs will be considered and included in the Bayesian Logistic Regression Model (BLRM).
Phase I (Group A and Group B): Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Phase I (Group A and Group B): Number of Participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Phase I (Group A and Group B): Dose Intensity | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized by means of descriptive statistics
Phase I (Group A and Group B): Duration of exposure to each study drug | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Duration of exposure (in months) to each study drug will be summarized by means of descriptive statistics
Phase II (Group A): Biochemical Response Rate (BCR) | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Biochemical Response Rate (BCR) is defined as prostate-specific antigen (PSA) decline to < 0.2 ng/mL at 6 months, confirmed by a second PSA measurement ≥ 3 weeks later.

SECONDARY OUTCOMES:
Phase I (Group A): Plasma concentrations of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Tulmimetostat and Darolutamide pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase I (Group A): AUC of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) and Area under the concentration-time curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) will be listed and summarized using descriptive statistics.
Phase I (Group A): Cmax of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Phase I (Group B): Plasma concentrations of Tulmimetostat and Abiraterone | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Day 2 (0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Tulmimetostat and Abiraterone pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase I (Group B): AUC of Tulmimetostat and Abiraterone | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Day 2 (0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) and Area under the concentration-time curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) will be listed and summarized using descriptive statistics.
Phase I (Group B): Cmax of Tulmimetostat and Abiraterone | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours), Day 2 (0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Phase II (Group A): Radiographic progression free survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 79 months
  Radiographic progression free survival (rPFS) is defined as the time between randomization and the first occurrence of disease progression as per PCWG3-modified RECIST v1.1 or death due to any cause
Phase II (Group A):Overall survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 79 months
  Overall survival (OS) is defined as the time between randomization to date of death due to any cause
Phase II (Group A): Objective response (OR) | From date of randomization until date of confirmed Complete Response (CR) or Partial Response (PR), assessed up to approximately 79 months
  Objective response (OR) is defined as a confirmed Complete Response (CR) or Partial Response (PR) per Prostate Cancer Working Group 3 (PCWG3)-modified RECIST 1.1 as assessed by the Investigator
Phase II (Group A): Best Overall response (BOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 79 months
  Best Overall response (BOR) is defined as the best response per PCWG3-modified RECIST 1.1 as assessed by the Investigator from the start of the treatment until disease progression/recurrence
Phase II (Group A): Duration of response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 79 months
  Duration of response (DOR) defined as time between first documented CR/PR and disease progression per PCWG3-modified RECIST 1.1 as assessed by the Investigator or death due to any cause
Phase II (Group A): Prostate-Specific Antigen 50 (PSA50) | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Prostate-Specific Antigen 50 (PSA50) is defined as a ≥ 50% decrease in PSA levels from baseline at any timepoint, confirmed by a second PSA measurement ≥ 3 weeks without any PSA progression in between
Phase II (Group A): Biochemical Response of <0.1 ng/mL | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Biochemical Response of <0.1 ng/mL is defined as PSA level < 0.1 ng/mL at any timepoint during the trial from randomization
Phase II (Group A): Time to castration-resistant prostate cancer (CRPC) | From date of randomization until date of PSA progression, radiological progression by bone lesions, or radiological progression by soft tissue and visceral lesions, whichever comes first, assessed up to approximately 79 months
  Time to castration-resistant prostate cancer (CRPC) is defined as the time from randomization to the first occurrence of one of the following events: PSA progression, radiological progression by bone lesions, or radiological progression by soft tissue and visceral lesions
Phase II (Group A): Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Phase II (Group A): Number of Participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Phase II (Group A): Dose Intensity | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized by means of descriptive statistics
Phase II (Group A): Duration of exposure to each study drug | From date of randomization till 30 days safety fup, assessed up to approximately 79 months
  Duration of exposure to each study drug will be summarized by means of descriptive statistics
Phase II (Group A): Plasma concentrations of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  In selected number of participants receiving Tulmimetostat and Darolutamide combination therapy in Phase II, or in selected number of participants if only one dose level of Tulmimetostat is evaluated in combination with Darolutamide in Phase II, Tulmimetostat and Darolutamide pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase II (Group A): AUC of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  In selected number of participants receiving tulmimetostat and darolutamide combination therapy in Phase II, or in selected number of participants if only one dose level of tulmimetostat is evaluated in combination with darolutamide in Phase II, venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) and Area under the concentration-time curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) will be listed and summarized using descriptive statistics.
Phase II (Group A): Cmax of Tulmimetostat and Darolutamide | Cycle 1-2: Day 1 (0 hour, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours). Cycle 1: Day 2 (Tulmimetostat only: 0 hour and 24 hours), Days 8 and 15 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  In selected number of participants receiving tulmimetostat and darolutamide combination therapy in Phase II, or in selected number of participants if only one dose level of tulmimetostat is evaluated in combination with darolutamide in Phase II, venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Phase II (Group A): Plasma concentrations of Tulmimetostat | Cycle 1-2: Day 1 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Tulmimetostat pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels by treatment arms
Phase II (Group A): AUC of Tulmimetostat | Cycle 1-2: Day 1 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) and Area under the concentration-time curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) will be listed and summarized using descriptive statistics.
Phase II (Group A): Cmax of Tulmimetostat | Cycle 1-2: Day 1 (0 hour and 2 hours). Cycles 3-5: Day 1 (0 hour). 1 cycle = 28 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Phase II (Group A): Time to first symptomatic skeletal event (TTSSE) | From randomization until the first occurrence of a new symptomatic bone fracture, spinal cord compression, tumor-related orthopedic surgery, radiation therapy for bone pain, or death, assessed up to 79 months.
  Time to first symptomatic skeletal event (TTSSE) is defined as the time from randomization to the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (2):
  - Wichita Urology Group PA, Wichita, Kansas
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Novartis Investigative Site, Wollongong, New South Wales, Australia
- Novartis Investigative Site, Guangzhou, China
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com